CLINICAL TRIAL: NCT03183544
Title: Kinetics, Biodistribution, Dosimetry and Safety Phase 1 Study With 68Ga-PSMA-11 Sterile Cold Kit, in Healthy Male Volunteers and Patients With Limited Recurrent Prostate Cancer
Brief Title: Dosimetry and Safety Phase 1 Study With 68Ga-PSMA-11 Sterile Cold Kit
Acronym: PSMA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017/30MAI/305
Record Dates: First submitted 2017-06-01; First posted 2017-06-12 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Prostatic Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: 5 patients with limited recurrent prostate cancer and 3 healthy volunteers will be enrolled in this clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gallium-68 PSMA-11 prepared using PSMA-11 Sterile Cold Kit (Experimental): Single injection for diagnostic use only
  Interventions: Combination Product: Gallium-68 PSMA-11 prepared using PSMA-11 Sterile Cold Kit

INTERVENTIONS:
Combination Product: Gallium-68 PSMA-11 prepared using PSMA-11 Sterile Cold Kit — The patients will receive a single injection of Gallium-68 PSMA-11 to diagnose biochemical relapse of prostate cancer after treatment.

SUMMARY:
Prostate cancer is the most common cancer in men. Early detection of primary diseases and recurrence is crucial for patient counseling and management. Conventional imaging modalities (CT-MRI) are limited to detect recurrence.

Choline-based PET/CT is currently widely used as primary staging tool in prostate cancer and in patients with suspicious recurrent disease.

Compared to choline-based tracers, 68Ga-PSMA ligands have been shown to have a higher diagnostic efficacy and to increase the detection of metastases even at low PSA levels. The most widely used prostate-specific membrane antigen (PSMA) ligand is PSMA-11. A supplier, ANMI, has developed a kit formulation of PSMA-11 which will be test in this clinical trial.

DETAILED DESCRIPTION:
Prostate cancer represents the most common cancer in men and accounts for the third most common cancer death in men. Up to 50% of all patients undergoing radical prostatectomy or radiotherapy for primary treatment of prostate cancer develop biochemical recurrence. Early detection of primary diseases and recurrence is crucial for patient counseling and management. Conventional imaging modalities such as computed tomography (CT) or magnetic resonance imaging (MRI) are limited because they focus on morphologic information such as lymph node size and tissue structure.

Positron emission tomography/computed tomography (PET/CT) is a hybrid imaging technique combining functional and morphological information. Choline-based PET/CT is currently widely used as primary staging tool in prostate cancer and in patients with suspicious recurrent disease. Compared to choline-based tracers, 68Ga-PSMA ligands have been shown to have a higher diagnostic efficacy and to increase the detection of metastases even at low PSA levels. The most widely used prostate-specific membrane antigen (PSMA) ligand is PSMA-11. A supplier, ANMI, has developed a kit formulation of PSMA-11 which can be labeled at room temperature by direct incubation of the kit with the gallium-68 eluted from a 68Ge/68Ga generator.

ELIGIBILITY:
Inclusion Criteria:

* For all individuals

  * Male gender
  * Normal renal function (MDRD glomerular filtration rate >60/ml/min/1.73m2)
  * Normal liver function (bilirubin, alanine aminotransferase [ALT], aspartate aminotransferase [AST] and gamma glutamyltransferase [GGT] <2x upper limit of normal [ULN]
  * Normal bone marrow function (hemoglobin [Hb]>12g/dl, white blood cells [WBC]>4500/µl, platelets>140,000/µl)
  * Informed consent For patients with limited recurrent prostate cancer
  * ≥18 years of age
  * Radical therapy by surgery or radiotherapy
  * Prostate specific antigen [PSA] level between 0.5 and 2ng/ml confirmed within two weeks before inclusion
  * Negative or inconclusive findings with standard imaging techniques as assessed by the referring physician with e.g. thoraco-abdominal Computed Tomography [CT] scan, bone scan or Magnetic Resonance Imaging [MRI] within the previous two months before inclusion
  * Ability to undergo a one-day experimental study and the appropriate follow-up For healthy volunteers
  * 18 - 70 years of age
  * No known prostate disease according to medical history, current symptoms and digital rectal examination
  * PSA level <3ng/ml
  * Ability to undergo a two-day experimental study within a time interval of 7-15 days and the appropriate follow-up.

Exclusion Criteria:

* For all individuals

  * Urinary incontinence
  * Chronic renal disease (except nephroangiosclerosis or early diabetic nephropathy) even if renal function is normal
  * Concomitant malignant disease or diagnosis of cancer within five years prior to enrollment (except basal cell carcinoma)
  * History of salivary gland disease (except recovered childhood mumps)
  * History of surgery or radiotherapy of the salivary gland or neck
  * Medical or psychiatric condition that would preclude the conduct of the study to its end
  * Pregnant partner

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This protocol concerns only patients with prostatic cancer and male healthy volunteers.
Enrollment: 3 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma concentration | at day 0
  Measures based on blood tests
Maximum Urine concentration | Up to 6 months
  Based on urine samples

SECONDARY OUTCOMES:
Time dependant changes of the injected activity per organ | at day 0
  Calculation of mean organ-absorbed doses and effective doses
Incidence of treatment emergent adverse events | Up to 6 months
  Vital signs, laboratory parameters and adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: François Jamar, MD, PhD, Study Director — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD at this moment